CLINICAL TRIAL: NCT05322525
Title: A Research Study to Evaluate the Safety and Potential Efficacy of ON101 Cream for the Treatment of Venous Leg Ulcers.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the product development strategy adjustment, the Sponsor terminated this study.
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ON101CLAS03
Record Dates: First submitted 2021-03-22; First posted 2022-04-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Venous Leg Ulcers (VLU)
Keywords: ON101; Fespixon; Venous leg ulcers; C6 or C6R

STUDY DESIGN:
Intervention Model Description: The study consists of 3 periods, a Screening/Run-in period, a treatment period, and a follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ON101 Cream (Experimental): Single arm of VLU group for ON101 Cream
  Test drug:
  1. Name: ON101
  2. Dosage form: Topical cream
  3. Active ingredients: Extracts of Plectranthus amboinicus and Centella Asiatica
  4. Dose(s): Apply 1 cc per 5 cm2 ulcer size (not exceeding 2 mm in thickness)
  5. Dosing schedule: Apply once a day
  Interventions: Drug: ON101 Cream

INTERVENTIONS:
Drug: ON101 Cream — Test drug:
  1. Name: ON101
  2. Dosage form: Topical cream
  3. Active ingredients: Extracts of Plectranthus amboinicus and Centella Asiatica
  4. Dose(s): Apply 1 cc per 5 cm2 ulcer size (not exceeding 2 mm in thickness)
  5. Dosing schedule: Apply once a day
  Other Names: Fespixon

SUMMARY:
A Research Study to evaluate the safety and potential efficacy of ON101 cream for the treatment of venous leg ulcers.The objectives of the study are to determine the safety and to explore the potential efficacy of ON101 cream in patients with venous leg ulcers.

DETAILED DESCRIPTION:
This is a multi-center, open-label study to investigate the Safety and Potential Efficacy of ON101 Cream in Venous Leg Ulcers (VLU) patients. Subjects with VLU of CEAP C6 (active venous ulcer) or C6R (recurrent active venous ulcer) are to be included in this study. If a subject has more than one ulcer on the leg, the most severe ulcer then the largest ulcer that confirm to meet the eligibility criteria will be selected for study evaluation.

12 eligible subjects will be enrolled and receive ON101 cream treatment. Enrolled subjects will be instructed to apply the study treatment on the selected target ulcer for a maximum of 18 weeks, until the ulcer complete closure (ulcer size of 0) for two consecutive visits that at least 2 weeks apart, or until the subject exit the study prematurely due to any reason. Identical standard of care (SoC) procedure will be performed in both the control and investigational product arms throughout the study period, which including ulcer cleansing, debridement if necessary, and application of a suitable dressing and compression system until complete ulcer closure. Subjects are required to apply compression device at least 8 hours per day throughout the treatment period.

The study consists of three periods, a 2-week Screening/Run-in period, an up-to-18-week Treatment period, and a 1-to-2-week Follow-up period. The Screening/Run-in period is to ensure the subjects' eligibility and their compliance to compression therapy and to exclude subjects who demonstrate substantial healing resulting solely from improved compliance with SoC. The Treatment period is to determine the safety and to explore the potential efficacy of the study product. The Follow-up period is to assess the safety. During the Follow-up period, SoC will be provided to subjects with non-healing or recurrent target ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed a written informed consent prior to the study procedure
2. Male or female aged at least 20 years old
3. Venous outflow/venous capacitance (VO/VC) compatible with venous insufficiency measured at screening visit or within 3 months prior to enrollment
4. Has adequate vascular perfusion of the affected limb, confirmed by Ankle-Brachial Index (ABI) ≥ 0.8 and ≤ 1.3 measured at screening visit or within 3 months prior to enrollment
5. The target ulcer have all of the following characteristics:

   1. C6 or C6R per the Clinical-Etiology-Anatomic-Pathophysiologic (CEAP) Classification System;
   2. Located between the knee and ankle (at or above the malleolus);
   3. No active infection;
   4. Post debridement ulcer area is ≥ 3 cm2 and ≤ 20 cm2 at the time of enrollment;
   5. Has been presented for at least 6 weeks before enrollment;
   6. A minimum of 2 cm margin between the qualified target ulcer and any other ulcers on the target limb (post debridement);
   7. Involves a full thickness skin loss, but without exposure of tendon, muscle, or bone;
   8. Must be nonhealing as defined as ≤ 30% reduction in ulcer area in response to standard of care (SoC) during the 2-week run-in period
6. Considered by the Investigator to be compliant/adhere to the compression device during the 2-week run-in period
7. If female of child-bearing potential, has a negative pregnancy test on urine at screening and must not be breastfeeding
8. Able and willing to attend the scheduled visits and comply with the study procedures.

Exclusion Criteria:

1. Presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement
2. With deep vein thrombosis within 4 weeks prior to enrollment
3. Has endovenous surgery planned or performed within 4 weeks prior to enrollment
4. Laboratory values at Screening of:

   1. Liver function test (total bilirubin, aspartate aminotransferase [AST], or alanine aminotransferase [ALT]) > 3x the upper limit of normal, or
   2. Poor nutritional status defined as albumin < 2.5 g/dL, or
   3. Renal function test (serum creatinine) > 2x the upper limit of normal, or
   4. Glycosylated hemoglobin (HbA1c) ≥ 9 %
5. Presence of any clinically significant medical condition(s) in medical history during screening period that, in the opinion of the Investigator, could interfere with ulcer healing, including but not limited to the following:

   1. Systemic infection not controlled by suitable antibiotic treatment
   2. Active malignant disease. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, maybe considered for study entry.
   3. Acquired immune deficiency syndrome (AIDS) or HIV positive
6. Has received treatment with immunosuppressive or chemotherapeutic agents, radiotherapy, or systemic corticosteroids within 4 weeks prior to enrollment
7. Heavy smoker (≥ 20 cigarettes per day)
8. Use of any investigational drug or therapy within 4 weeks prior to enrollment
9. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse problem, determined from the subject's medical history, which in the opinion of the Investigator, may pose a threat to subject compliance
10. Judged by the Investigator to be not suitable for study participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Safety endpoint(1) : Treatment-Emergent Adverse Event | Through study completion, an average of 6 months
  Incidence of treatment-emergent adverse event (TEAE); safety will be assessed by the incidence of adverse events, including overall AEs, AEs related to the ON101, study-ulcer-associated AEs and SAEs.
Safety endpoint(2-1) : Change from baseline in vital signs | Through study completion, an average of 6 months
  Incidence of treatment-emergent adverse event (AE) Change from baseline in vital signs:pulse rate(times/min), SBP/DBP(mmHg), Body Temperature (°C), and respiratory rate ( breaths/min)
Safety endpoint(2-2) : Change from baseline in physical examination | Through study completion, an average of 6 months
  Incidence of treatment-emergent adverse event (AE) Change from baseline in the physical examination: HEENT (head, eyes, ears, nose, and throat), mouth, skin, neck (including thyroid), lymph nodes, spine, cardiovascular system, respiratory system, gastrointestinal system, nervous system, musculoskeletal system, blood and blood-forming organs and mental status.
Safety endpoint(2-3) : Change from baseline in laboratory test | Through study completion, an average of 6 months
  Incidence of treatment-emergent adverse event (AE) Change from baseline in laboratory tests: Complete blood count (WBC, Neutrophils, Monocytes, Hb, MCV, MCH, MCHC, Platelet), Biochemistry (HbA1c, fasting blood glucose, triglyceride, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, total bilirubin, aspartate aminotransferase, alanine aminotransferase, creatinine, albumin), and Urinalysis (pH, protein, glucose, ketone, blood, urobilinogen, bilirubin, nitrite, leukocyte)

SECONDARY OUTCOMES:
Efficacy endpoint(1): ulcer healing time measured | Through study completion, an average of 6 months
  Time to complete ulcer healing:measured by the photo to ensure the target ulcer area, such as length, width,and depth changed
Efficacy endpoint(2): complete healing of the target ulcer | Through study completion, an average of 6 months
  Incidence of complete healing of the target ulcer:measured by the photo to ensure the target ulcer area, such as length, width,and depth changed.
Efficacy endpoint(3): change from baseline in the target ulcer area | Through study completion, an average of 6 months
  Mean change from baseline in the target ulcer area:measured by the photo to ensure the target ulcer area, such as length, width,and depth changed.
Efficacy endpoint(4): percentage change from baseline in the target ulcer area | Through study completion, an average of 6 months
  Percentage change from baseline in the target ulcer area:measured by the photo to ensure the target ulcer area, such as length, width,and depth changed
Efficacy endpoint(5): between target ulcer area and time to complete ulcer healing | Through study completion, an average of 6 months
  Correlation between target ulcer area and time to complete ulcer healing:measured by the photo to ensure the target ulcer area, such as length, width,and depth changed

CONTACTS AND LOCATIONS:
Overall Officials: Shyi-Gen Chen, MD, Study Director — Oneness Biotech Co., Ltd.
Locations (2):
- Taiwan (2):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
IIS study